CLINICAL TRIAL: NCT01661361
Title: Optimalisation of Therapeutic Drug Monitoring (TDM) of Vancomycin in Patients With Central Venous Port Devices
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Isabelle Spriet, PharmD, PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S54585
Record Dates: First submitted 2012-07-20; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Catheter-related Infection
Keywords: vancomycin; levels; central venous port device; peripherally obtained levels; dose adjustments; TDM
MeSH Terms: conditions — Catheter-Related Infections | interventions — Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vancomycin cohort
  Interventions: Procedure: blood levels

INTERVENTIONS:
Procedure: blood levels

SUMMARY:
Recently, it was reported that when vancomycin levels are determined after port sampling, levels can be falsely increased potentially leading to wrong dose adjustments.

The investigators conducted an in vitro experiment using several central venous port devices, in which different flushing techniques were evaluated yielding residual vancomycin levels of less than 0.5 mg/L.

In this study, the investigators want to evaluate this flushing technique in vivo in 15 patients admitted with catheter-related infection and treated with systemic vancomycin and vancomycin antibiotic lock.

The purpose is to assess if correct flushing can avoid spurious vancomycin levels obtained via port sampling.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* having central venous port device,
* treated with systemic vancomycin in combination with vancomycin antibiotic lock

Exclusion Criteria:

* pregnant women,
* children,
* patients with 'do not resuscitate' (DNR) code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted for catheter related infection with methicillin-resistant coagulase-negative staphylococci (MR-CNS) and treated with systemic vancomycin in combination with vancomycin antibiotic lock via central venous port device.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
comparison of central (via port device) and peripherally obtained vancomycin levels: the difference, when using the new flushing technique, is allowed to be maximally 0.5 mg/L | central and peripheral vancomycin levels will be obtained during steady state: this means starting from the 4th dose (= day 2) of vancomycin treatment. Vancomycin is usually given during 14 days after the last positive blood culture.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Principal Investigator — Pharmacy Dpt, University Hospitals Leuven; Jan Verhaegen, MD PhD, Study Chair — Medical Diagnostic Sciences, University Hospitals Leuven; Hans Prenen, MD PhD, Study Chair — Digestive ONcology, University Hosptials Leuven; Willy Peetermans, MD PhD, Study Chair — Internal Medicine, University Hospitals Leuven; Ludo Willems, PharmD PhD, Study Chair — Pharmacy Dpt., University Hosptials Leuven